CLINICAL TRIAL: NCT02105441
Title: Cochlear Implantation Among Adults and Older Children With Unilateral or Asymmetric Hearing Loss
Acronym: CI and SSD
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew L. Carlson, M.D., Associate Professor of Neurosurgery and Otolaryngology, Mayo Clinic
Other Study IDs: 13-009050
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Severe Unilateral Sensorineural Hearing Loss
Keywords: cochlear implant
MeSH Terms: interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cochlear implant: How well patients with cochlear implants understand speech in noise with implant on, compared to implant off.
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Implantable hearing device

SUMMARY:
Do adults and children over 7 years of age with unilateral or assymetric hearing loss benefit from cochlear implantation on the worst hearing side.

DETAILED DESCRIPTION:
Unilateral hearing loss is known to impair binaural hearing abilities. Specifically, localization, speech understanding in noise, and binaural squelch suffer due to lack of binaural timing and level cues. This study is designed to examine how binaural hearing is improved following cochlear implantation on the impaired side. The study endpoints are collected at 6 months and 12 months post activation of the implant.

This is not a funded study. All costs are billed through insurance for reimbursement. There is an insurance approval process that we move through after a participant has been evaluated at the Mayo Clinic and found to be a candidate for cochlear implantation.

ELIGIBILITY:
Adults

* 18 years of age or older,
* Hearing loss in the ear to be implanted must such that speech understanding is not possible with a well fitted hearing aid. Specifically, less than 40% monosyllabic word understanding when that ear is tested in the best-aided condition and the other ear is sufficiently occluded or masked.
* Onset of hearing loss in the adult group must be post-lingual (after three years of age)

Children

* Children 7 years of age and older
* Hearing loss in the ear to be implanted configured such that word understanding is less 40% in the best aided condition
* Onset of hearing loss in the pediatric group must be post-lingual (after three years of age)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes adults and children over 7 years of age who have suffered single sided deafness. Word understanding on the impaired side must not exceed 50% correct in the best aided condition.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Listening Effort | one year post operative test time
  A dual task performance paradigm will be used in which both the primary task and the secondary task will be performed simultaneously. The primary task will consist of speech recognition testing in varying levels of background noise and quiet, whereas the secondary task will consist of a motor reaction to a randomly presented light

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Carlson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States